CLINICAL TRIAL: NCT05963880
Title: Concordance Between Central Blood PRessure dEvices In Nephrology Patients (CBP-REIN)
Brief Title: Concordance Between Central Blood PRessure dEvices In Nephrology Patients
Acronym: CBP-REIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding to enroll all planned participants
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CBP-REIN
Record Dates: First submitted 2023-05-12; First posted 2023-07-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Chronic Kidney Disease; Blood Pressure
Keywords: central blood pressure
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — Sphygmomanometers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Advanced CKD group (Experimental): Patients with eGFR < 30 ml/min/1.73m2 not on dialysis
  Interventions: Device: Brachial and Central BP measurements with Mobil-o-Graph NG device (IEM), WatchBP Office device (Microlife), BP+ device (Uscom) and Oscar 2 with SphygmoCor inside device (SunTech)
- Dialysis groups (Experimental): Patients on hemodialysis or peritoneal dialysis
  Interventions: Device: Brachial and Central BP measurements with Mobil-o-Graph NG device (IEM), WatchBP Office device (Microlife), BP+ device (Uscom) and Oscar 2 with SphygmoCor inside device (SunTech)
- Hypertension group (Experimental): Patients with BP > 135/85 mmHg or taking any antihypertensive medication with normal kidney function (eGFR > 60 ml/min/1.73m2)
  Interventions: Device: Brachial and Central BP measurements with Mobil-o-Graph NG device (IEM), WatchBP Office device (Microlife), BP+ device (Uscom) and Oscar 2 with SphygmoCor inside device (SunTech)
- Control group (Active Comparator): Normotensive patients without any antihypertensive drugs or chronic kidney disease
  Interventions: Device: Brachial and Central BP measurements with Mobil-o-Graph NG device (IEM), WatchBP Office device (Microlife), BP+ device (Uscom) and Oscar 2 with SphygmoCor inside device (SunTech)

INTERVENTIONS:
Device: Brachial and Central BP measurements with Mobil-o-Graph NG device (IEM), WatchBP Office device (Microlife), BP+ device (Uscom) and Oscar 2 with SphygmoCor inside device (SunTech) — All participants will have three readings at 1-min interval after a 5-min seated rest with each device. The order in which each device will be tested is randomized.

SUMMARY:
The most accurate way to determine intra-aortic BP is to obtain invasive measures by vascular catheterization, which is not possible to perform routinely during the regular follow-up of patients. However, in recent years, devices used to estimate central BP have been designed and approved for clinical use. These devices can determine aortic BP in a non-invasive way using various techniques and algorithms and offer a high degree of precision when compared to invasive measurements of intraaortic BP. On the other hand, certain characteristics specific to the different devices mean that the central BP values obtained may not be interchangeable. It is therefore important to determine the degree of agreement of central BP values obtained using commercially available devices.

This study aims to determine the degree of agreement between central BP measurements obtained using 4 devices commonly used to measure central blood pressure, i.e. Mobil-o-Graph NG (IEM, Germany), WatchBP Office (Microlife, Taiwan), Oscar 2 with SphygmoCor inside (SunTech, USA) and BP+ (Uscom, Australia). These four devices record the shape of the pulsatile wave and then derive the central BP using an algorithm. The main differences between these devices lie in this algorithm, or "transfer function,", which is unique to each and the calibration used. All use a brachial cuff to capture the pulse waveform and can easily be used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- Age 18-80 years old

Exclusion Criteria:

* Ongoing atrial fibrillation
* Arm circumference incompatible with the blood pressure cuffs for all devices (<18 cm or > 50 cm)
* Incapacity to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Central SBP difference | at enrollment (time 0)
  Differences in the central SBP measured by each device

SECONDARY OUTCOMES:
Brachial SBP difference | at enrollment (time 0)
  Differences in the brachial cuff SBP measured by each device
Central DBP difference | at enrollment (time 0)
  Differences in the central DBP measured by each device
Brachial DBP difference | at enrollment (time 0)
  Differences in the brachial cuff DBP measured by each device

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada